CLINICAL TRIAL: NCT01681368
Title: Phase II Open Label Non-Randomized Single Agent Study of the SMAC (Second Mitochondrial-Derived Activator of Caspases)-Mimetic Birinapant (TL32711; NSC 756502) in Relapsed Platinum Resistant or Refractory Epithelial Ovarian Cancer, Primary Peritoneal
Brief Title: Birinapant for Advanced Ovarian, Fallopian Tube, and Peritoneal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Accrual was terminated for lack of a clinical benefit.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Christina Annunziata, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 120191; 12-C-0191
Record Dates: First submitted 2012-09-05; First posted 2012-09-07 (Estimated); Results first posted 2015-02-03 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Epithelial Ovarian Cancer; Peritoneal Neoplasms; Fallopian Tube Neoplasms
Keywords: NF-Kappa B Pathway; Response Biomarkers; Progression-Free Survival; Pharmacokinetics; Pharmacodynamics
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Peritoneal Neoplasms; Fallopian Tube Neoplasms | interventions — birinapant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Birinapant for Advanced Ovarian,Fallopian Tube & Peritoneal Ca (Experimental): single arm
  Interventions: Drug: Birinapant (TL32711)

INTERVENTIONS:
Drug: Birinapant (TL32711) — 47mg/m^2 intravenous (IV) on days 1, 8 and 15 of each 28 day cycle

SUMMARY:
Background:

- Birinapant is an experimental cancer treatment drug. It removes certain proteins in cells, which helps to kill the cells. The drug is more likely to cause the death of cancer cells than normal cells because cancer cells have more of these proteins. Studies suggest that it can help treat ovarian cancer, primary peritoneal cancer, or fallopian tube cancer. Researchers want to see how well Birinapant works against the three types of cancer.

Objectives:

- To test the effectiveness of Birinapant for ovarian, primary peritoneal, or fallopian tube cancer.

Eligibility:

- Women at least 18 years of age who have ovarian, primary peritoneal, or fallopian tube cancer that has not responded to standard treatment.

Design:

* Participants will be screened with a physical exam and medical history. Blood and urine samples will also be collected. Tumor tissue samples may be collected before treatment. Imaging studies will also be performed.
* Participants will have an infusion of Birinapant once per week for 3 weeks in a row, followed by a break for a week on the fourth week. This 4-week schedule is one cycle of treatment.
* Treatment will be monitored with frequent blood tests and imaging studies.
* Another optional tumor biopsy will be collected 6 weeks after the start of treatment.
* Treatment will continue as long as the cancer does not grow and the side effects are not severe.

DETAILED DESCRIPTION:
BACKGROUND:

* Ovarian cancer is the ninth most common cancer in women (excluding skin cancer). It ranks fifth as the cause of cancer death in women. In the United States, 21,550 new cases and 14,600 deaths are estimated annually.
* Approximately 90% of primary malignant ovarian tumors are epithelial (carcinomas).
* Although over 70% of women with advanced disease respond to optimal debulking surgery followed by platinum-taxane based chemotherapy, duration of response is short and relapse is common. Subsequent responses to salvage therapy regimens tend to be brief (less than six months) due to the tumors progressive resistance to chemotherapy(1).
* A family of proteins, known as the Inhibitors of Apoptotic Proteins (or IAPs), plays a critical role in blocking the apoptotic signals at multiple points. IAPs regulate a number of pathways including classical or alternative nuclear factor-kappa B (NF-(K)B) function, and activation of apoptosis through either the extrinsic or intrinsic pathway. Baculoviral IAP repeat-containing protein 1 (cIAP1) acts as a critical switch to promote the pro-survival nuclear factor kappa-B (NF-B) pathway and prevent caspase activation.
* In normal cells that are stimulated to undergo apoptosis by either the extrinsic or intrinsic pathway, second mitochondrial-derived activation of caspares (SMAC) is released from the mitochondria, which antagonizes IAP, removes blockade to activated caspase function, and thereby enables apoptotic cell death. In tumor cells, however, apoptosis is dysregulated due to insufficient amounts of SMAC or upstream blockades to apoptotic activation.
* Classical activation of NF-(K)B is dependent on the presence of cIAP1 and cIAP2 proteins as part of the TNF receptor-associated factor 2 (TRAF2) complex. SMAC inhibits cIAP1 and cIAP2, leading to inactivation of tumor necrosis factor alpha (TNFalpha) mediated NF- B activation. SMAC inhibition of cIAP1 and cIAP2 leads to pathway up-regulation. Birinapant (TL32711) is a synthetic peptidomimetic antagonist of IAPs (a SMAC-mimetic), which mimics endogenous SMAC resulting in the rapid and irreversible initiation of apoptotic cell death. SMAC-mimetics represent a novel targeted therapeutic approach for cancer therapy. The addition of a SMAC mimetic, can inhibit NF- B activity, down-regulate cell survival pathways, and overcome blockades to the apoptotic pathway leading to increased tumor cell death.
* Our laboratory has demonstrated that serous ovarian cancers have cell-autonomous activation of NF-B signaling which was shown to correlate with poor prognosis.
* Therefore, we hypothesize that the SMAC-mimetic activity of birinapant may be selectively toxic to those ovarian cancers that display high canonical NF-(K)B activity.
* To summarize, relapsed platinum refractory or resistant ovarian cancer is a disease with limited therapeutic options and poor prognosis. Birinapant offers the opportunity to develop an effective and well tolerated therapeutic for the significant unmet need.

OBJECTIVES:

* The primary objective is to determine the efficacy as defined by Gynecologic Oncology Group (GOG) criteria2 as either objective response or progession-free survival lasting greater than 6 months, in patients with relapsed platinum refractory or resistant ovarian cancer, primary peritoneal cancer, fallopian tube cancer treated with birinapant.
* The seconday objectives include overall survival, safety and tolerability of single agent birinapant in this population.

ELIGIBILITY CRITERIA:

* Females greater than or equal to 18 years of age with histologically proven advanced metastatic or unresectable epithelial ovarian cancer that is relapsed or refractory to prior platinum-based standard care systemic regimen.
* Life expectancy greater than 3 months.
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2.
* Adequate organ functionas defined by liver, kidney, and hematologic laboratory testing.

Design:

* This is an open label, non-randomized phase II trial to determine the efficacy of administration of the SMAC-mimetic birinapant in patients with relapsed platinum refractory or resistant ovarian cancer, primary peritoneal cancer, fallopian tube cancer.
* Birinapant will be given as a single agent until disease progression once weekly for three weeks of 4 week intervals.
* The primary endpoint will be efficacy defined according to the GOG guidelines as overall response rate or progression-free survival lasting at least 6 months. Overall survival, toxicity and modulation of signal events in tumor are secondary measures.
* Patients will be evaluated at baseline and prior to each cycle by history and physical examination and every two cycles by examination and imaging studies (computed tomography (CT) scan). Laboratory studies will be performed weekly prior to each dose except on week 4 (rest week).
* Tumor biopsy will be performed prior to birinapant initiation and an optional tumor biopsy will be performed 2 to 48 hours after cycle 2 day 15 infusion.
* Peripheral blood mononuclear cells will also be harvested at the same time points as the biopsies.
* Reassessment imaging (computed tomography (CT) scan) to document response will be performed at the end of 2 cycles and every 2 cycles thereafter.

ELIGIBILITY:
* INCLUSION CRITERIA:

Study participants will be eligible for study participation if they are/have:

* Females greater than or equal to 18 years of age. Because no dosing or adverse event data are currently available on the use of birinapant in patients < 18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.
* Able to understand and voluntarily sign a written informed consent, and are willing and able to comply with the protocol requirements including the requirement for biopsies for research purposes.
* Advanced metastatic or unresectable epithelial ovarian cancer, primary peritoneal cancer or fallopian tube cancer that is relapsed and resistant or refractory to prior platinum-based standard care systemic regimen. Patients who are unable to receive further platinum, due to either allergic reaction or other medical reason, are eligible for the protocol. There is no limitation on the amount of prior therapies allowed.
* Patients must be at least 4 weeks from previous therapy (chemotherapy, hormonal therapy, and radiation therapy, immunotherapy and monoclonal antibodies, alternative therapy or investigational therapeutic agents). Patients who have had cranial radiation therapy need to have completed it greater than or equal to 8 weeks prior to commencing on study. Patients are permitted to receive investigational imaging agents while on study.
* Patients who have had major surgery must be fully recovered and require a recovery period of greater than or equal to 4 weeks prior to enrolling on study.
* Histopathologic diagnosis must be confirmed in the Laboratory of Pathology (LP), National Cancer Institute (NCI).

A block of the primary tumor, or access to recut slides is preferred. If this is unavailable, a recent resection specimen of a metastatic site is required for entry. In addition, access to archival formalin fixed paraffin embedded (FFPE) tumor blocks will be requested to perform correlative studies. Study participants with the following histologic epithelial ovarian cancer cell types are eligible: Serous adenocarcinoma, endometrioid adenocarcinoma, mucinous adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma, transitional cell carcinoma, malignant Brenner's Tumor, or adenocarcinoma not otherwise specified (N.O.S).

* Patients must have measurable disease by Response Evaluation Criteria in Solid Tumors defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as greater than or equal to 20 mm with conventional techniques or as greater than or equal to 10 mm with spiral computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam and a sentinel lesion adequate for core biopsy through percutaneous biopsy. See Section 13 for the evaluation of measurable disease.
* Life expectancy greater than 3 months.
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to less than or equal to 2.
* Adequate renal function, defined as serum creatinine less than or equal to 1.5 X upper limit of normal (ULN), or measured creatinine clearance greater than or equal to 60 ml/min/1.73m^2.
* Adequate hepatic function, defined as aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels less than or equal to 3 X ULN and total bilirubin < 1.5 X ULN, unless known diagnosis of Gilberts syndrome.
* Adequate bone marrow function, defined as absolute neutrophil (ANC) greater than or equal to 1,500/mm^3 (greater than or equal to1.5 X10^6/L), platelet count greater than or equal to 75,000/mm^3 (greater than or equal to 75 X10^6/L), and hemoglobin greater than or equal to 10 mg/dL (transfusion to obtain hemoglobin greater than or equal to 10 mg/dL within 24 hours prior to dosing is allowed).
* Contraception is not a consideration as these patients have all had surgical removal of their reproductive organs. Pregnant women are excluded from this study because birinapant may have potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with birinapant, breastfeeding should be discontinued prior to enrollment.

EXCLUSION CRITERIA:

1. Known or suspected diagnosis of human immunodeficiency virus or chronic active hepatitis B or C. Viral testing is not required. The reason for exclusion is insufficient evidence demonstrating safety of administration of birinapant in patients with human immunodeficiency virus (HIV), hepatitis B or C due to theoretical risk of unmasking or exacerbating these serious viral illnesses since birinapant may impair immunological function. Data are not currently available on risk of interaction with antiretroviral drugs. HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with birinapant. The potential immune suppressive effects and T-cell depletion associated with birinapant pose an additional increased risk to these patients. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
2. Symptomatic or uncontrolled brain metastases requiring current treatment (< 8 weeks from last cranial radiation or < 4 weeks from last steroids). (Patients with abnormal clinical exam or history will require a head CT or MRI to rule out or confirm brain metastases).
3. Impaired cardiac function or clinically significant cardiac disease including the following:

   1. New York Heart Association grade III or IV congestive heart failure.
   2. Myocardial infarction within the last 12 months prior to dosing with birinapant.
   3. Subjects known to have impaired left ventricular ejection fraction (LVEF) according to institutional standards must be excluded.
4. Lack of recovery of prior adverse events to Grade less than or equal to1 severity (National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] v 4.03) (except alopecia) due to therapy administered prior to the initiation of study drug dosing. Stable persistent grade 2 peripheral neuropathy may be allowed as determined on a case-by-case basis at the discretion of the Investigator as birinapant has not been shown to cause or exacerbate peripheral neuropathy.
5. Known allergy to any of the formulation components of birinapant including citric acid monohydrate, sodium citrate dehydrate, and sodium chloride.
6. Any concurrent disease and/or medical condition that in the opinion of the Investigator would prevent the subjects participation, render the subject at excessive risk or limit the subjects compliance with the protocols required evaluations.
7. Patients with active infection will not be eligible, but may become eligible once infection has resolved and they are at least 7 days from completion of antibiotics.
8. Another previous or current malignancy within the last 5 years, with the exception of non-melanoma skin cancer, cervical carcinoma in situ curatively treated, ductal or lobular carcinoma in situ curatively treated and without ongoing therapeutic intervention. Patients with breast cancer (BRCA) 1 or 2 mutation, who have had a previous diagnosis of breast cancer are eligible if the breast cancer was diagnosed 5 years previously and distant or local recurrence of breast cancer has been outruled.
9. Concomitant chronic (daily or almost daily for greater than or equal to1 month prior) use of steroids or non-steroidal anti-inflammatory drugs (NSAIDS). Intermittent use of steroids as pre-medications is allowed. Based on research to date the tumor and tumor microenvironment production of tumor necrosis factor (TNF) alpha could promote anti-tumor activity. Theoretically, anti-inflammatories could blunt local production, limiting this possibly positive cofactor.
10. No concomitant use of complementary or alternative medication or other agents (investigational therapeutic agents) will be allowed without approval of a principal investigator (PI) or associate investigator (AI). Every effort will be made to maximize patient safety and minimize changes in chronic medications.
11. Patients with a recent history (within last 5 years) of autoimmune disease or inflammatory diseases will be excluded, for example, active rheumatoid arthritis,active inflammatory bowel disease or any chronic inflammatory conditions because birinapant synergizes with TNF in vitro.

INCLUSION OF MINORITIES:

Women from all racial/ethnic groups are eligible for this study if they meet the eligibility criteria.

To date, there is no information that suggests that differences in drug metabolism or disease response would be expected in one group compared to another. Efforts will be made to extend accrual to a representative population, but in this preliminary study, a balance must be struck between patient safety considerations and limitations on the number of individuals exposed to potentially toxic and/or ineffective treatments on the one hand and the need to explore ethnic aspects of clinical research on the other hand. If differences in outcome that correlate to ethnic identity are noted, accrual may be expanded or a follow-up study may be written to investigate those differences more fully. This study will be recruited through internal referral, our local physician referral base, and through Cancer Hotline information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 11 (Actual)
Dates: Start 2012-08-15 (Actual); Primary Completion 2013-12-09 (Actual); Study Completion 2014-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina M Annunziata, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaye SB. Management of platinum-sensitive relapsed ovarian cancer, with particular reference to the International Collaboration in Ovarian Neoplasm-4/Arbeitsgemeinschaft Gynakologische Onkologie Ovarian Cancer-2.2 trial. Int J Gynecol Cancer. 2005 May-Jun;15 Suppl 1:31-5. doi: 10.1111/j.1525-1438.2005.15354.x. PMID 15839956
- [Background] Rose PG, Tian C, Bookman MA. Assessment of tumor response as a surrogate endpoint of survival in recurrent/platinum-resistant ovarian carcinoma: a Gynecologic Oncology Group study. Gynecol Oncol. 2010 May;117(2):324-9. doi: 10.1016/j.ygyno.2010.01.040. Epub 2010 Feb 24. PMID 20185168
- [Background] Gordon AN, Granai CO, Rose PG, Hainsworth J, Lopez A, Weissman C, Rosales R, Sharpington T. Phase II study of liposomal doxorubicin in platinum- and paclitaxel-refractory epithelial ovarian cancer. J Clin Oncol. 2000 Sep;18(17):3093-100. doi: 10.1200/JCO.2000.18.17.3093. PMID 10963637
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-C-0191.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Birinapant for Advanced Ovarian,Fallopian Tube & Peritoneal Ca
Started | 11
Completed | 9
Not Completed | 2
Not completed — Refused further treatment | 1
Not completed — Refused further follow up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Birinapant for Advanced Ovarian,Fallopian Tube & Peritoneal Ca
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 2
Age, Continuous [Median (Standard Deviation); unit: years] | 58.87 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 11
Eastern Cooperative Oncology Group (ECOG) [Count of Participants; unit: Participants] — ECOG: 0 (Normal activity. Fully active, able to carry on all pre-disease performance without restriction.), 1 (Symptoms, but ambulatory. Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature (e.g., light housework, office work), and 2 (In bed <50% of the time. Ambulatory and capable of all self-care, but unable to carry out any work activities. Up and about more than 50% of waking hour.).
  Participants
    0 | 0
    1 | 10
    2 | 1
Histologic subtype, No. [Count of Participants; unit: Participants]
  Serous | 6
  Endometrioid | 1
  Clear cell | 1
  Classified | 3
No. of Prior Therapies [Count of Participants; unit: Participants]
  ≤3 | 1
  4-6 | 6
  ≥7 | 4
Type of Prior Therapy, No. [Number; unit: participants]
  Chemotherapy | 11
  Biologic | 6
  Hormonal | 5
  Vaccine | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response (Complete Response (CR) or Partial Response (PR) Defined by Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 Criteria) or Disease Stabilization for Greater Than 6 Months
Description: Per the RECIST criteria, CR is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10mm. Partial response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Birinapant for Advanced Ovarian,Fallopian Tube & Peritoneal Ca
Number analyzed (Participants) | 11
participants
  Complete Response | 0
  Partial Response | 0

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For a detailed list of adverse events, see the adverse event module.
Time Frame: 8 months
Measure: Number; unit: participants
Arm/Group | Birinapant for Advanced Ovarian,Fallopian Tube & Peritoneal Ca
Number analyzed (Participants) | 11
participants | 11

3. Secondary Outcome: Mean Plasma Concentration-Time Curve of Birinapant
Description: Measurement of the plasma concentration of the Birinapant over time. It is used to characterize drug absorption. The single values were analyzed with liquid chromatography/tandem mass spectrometry via a proprietary methodology (TetraLogic Pharma,Malvern, Pa). The values were grouped and averaged for each of the patients to obtain the mean value for each time point.
Time Frame: 30, 60, 120, 180 minutes after administration of first dose of Birinapant
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Birinapant for Advanced Ovarian,Fallopian Tube & Peritoneal Ca
Number analyzed (Participants) | 11
ng/mL
  Predose | 0 (0)
  30 minutes post end of infusion (EOI) | 699 (157)
  60 minutes post end of infusion (EOI) | 415 (84)
  120 minutes post end of infusion (EOI) | 202 (43)
  240 minutes post end of infusion (EOI) | 85 (20)

4. Secondary Outcome: Birinapant Concentration in Tumor Tissue
Description: Levels of Birinapant were measured in core needle biopsies of tumor that had been frozen at the time of acquisition.
Time Frame: Prior to treatment and 12 to 22 hours following Cycle 2 Day 15
Population: 4 patients did not have the second paired biopsy due to patient refusal.
Measure: Mean (Full Range); unit: ng/g
Arm/Group | Birinapant for Advanced Ovarian,Fallopian Tube & Peritoneal Ca
Number analyzed (Participants) | 7
ng/g | 952 [185 to 1830]

5. Secondary Outcome: Calculated Volume of Distribution of Birinapant at Steady State (Vss) in Tumor Tissue
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug.
Time Frame: 0-24hr
Measure: Mean (Full Range); unit: L
Arm/Group | Birinapant for Advanced Ovarian,Fallopian Tube & Peritoneal Ca
Number analyzed (Participants) | 11
L | 119 [80 to 183]

6. Secondary Outcome: Calculated Volume of Distribution of Birinapant at Steady State (Vss) in Plasma
Description: as for outcome 5
Time Frame: 0-24hr
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Birinapant for Advanced Ovarian,Fallopian Tube & Peritoneal Ca
Number analyzed (Participants) | 11
L | 132 (33)

7. Secondary Outcome: Ratio of Phosphorylated NF-kappaB-p65 Protein to Total NF-kappaBp65 Protein in Tumor Biopsy Samples
Description: Proteins were measured using capillary western blot and ratio was calculated between phosphorylated and total NF-kappaB p65. Core 1 tumor samples and peripheral blood mononuclear cells (PBMCs) from each time point were lysed in T-PER buffer (Thermo Scientific) for protein quantification by an automated capillary electrophoresis immunoassay system (Simple Western). The tumor protein lysate (40-60 ng) or PBMC protein lysate (16-77 ng) was analyzed according to the manufacturer's instructions (ProteinSimple, Santa Clara, Calif).
Time Frame: 0-6 weeks
Population: 4 patients refused second biopsy.
Measure: Mean (Full Range); unit: pixel intensity per ng protein
Arm/Group | Birinapant for Advanced Ovarian,Fallopian Tube & Peritoneal Ca
Number analyzed (Participants) | 7
pixel intensity per ng protein | 0.2 [0 to 0.4]

8. Secondary Outcome: Coexpression of Cleaved Caspase 3 and Gamma-H2AX in Fixed Specimens
Description: Tumor biopsies were measured for cleaved caspase 3 and gamma-H2A.X by immunofluorescence microscopy. Fold change was calculated by comparing the post-treatment measurements to the pre-treatment levels.
Time Frame: Pre treatment and post treatment of Birinapant, approximately 0-6 weeks
Population: Only 2 pairs of adequate pre- and post-treatment biopsy samples were available for analysis. The remaining paired samples were inadequate for immunohistochemistry because of necrotic debris in the post-treatment biopsy sample (1 specimen) or contamination with blood (4 specimens).
Measure: Median (Full Range); unit: Fold over baseline
Arm/Group | Birinapant for Advanced Ovarian,Fallopian Tube & Peritoneal Ca
Number analyzed (Participants) | 2
Fold over baseline | 3 [2 to 4]

9. Secondary Outcome: Total Clearance of Birinapant After Administration
Description: Clearance is a quantitative measure of the rate at which a drug substance is removed from the body.
Time Frame: 0-24hr
Measure: Mean (Full Range); unit: L/hr
Arm/Group | Birinapant for Advanced Ovarian,Fallopian Tube & Peritoneal Ca
Number analyzed (Participants) | 11
L/hr | 67.93091577 [45.1843727 to 105.7101965]

ADVERSE EVENTS:
Time Frame: 8 months
Arm/Group | Birinapant for Advanced Ovarian,Fallopian Tube & Peritoneal Ca
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 11/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Birinapant for Advanced Ovarian,Fallopian Tube & Peritoneal Ca (N=11)
Anemia (Blood and lymphatic system disorders) | 5 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Colonic obstruction (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Eye disorders - Other, specify (diplopia) (Eye disorders) | 1 (1)
Facial nerve disorder (Nervous system disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 6 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Birinapant for Advanced Ovarian,Fallopian Tube & Peritoneal Ca (N=11)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (4)
Alkaline phosphatase increased (Investigations) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 7 (10)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Anxiety (Psychiatric disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Chills (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Creatinine increased (Investigations) | 3 (4)
Diarrhea (Gastrointestinal disorders) | 5 (7)
Dizziness (Nervous system disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Edema trunk (General disorders) | 1 (1)
Fatigue (General disorders) | 5 (5)
Fever (General disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (3)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (3)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 (10)
Hypokalemia (Metabolism and nutrition disorders) | 2 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (4)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Lipase increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 4 (7)
Metabolism and nutrition disorders - Other, specify (low protein) (Metabolism and nutrition disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (6)
Platelet count decreased (Investigations) | 2 (3)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Serum amylase increased (Investigations) | 3 (4)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Weight loss (Investigations) | 2 (2)
White blood cell decreased (Investigations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No